CLINICAL TRIAL: NCT01568138
Title: This Study is a Multi-center, Prospective, Single-armed, Study Designed to Evaluate the Safety and Feasibility of the BioVentrix PliCath HF System for Left Ventricular (LV) Volume and Radius Reduction Through Scar Exclusion in Patients Whose Systolic HF is Due to Ischemic Cardiomyopathy.
Brief Title: Prospective Study of the BioVentrix PliCath HF™ System for the Treatment of Ischemic Cardiomyopathy
Acronym: CONFIGURE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioVentrix (Industry)
Collaborators: Ohio State University (Other); Centro Diagnostico Italiano (Unknown); Advance Research Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20032-P
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure
Keywords: Ventricular Remodeling
MeSH Terms: conditions — Heart Failure; Ventricular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: PliCath HF System — To evaluate the safety and feasibility of the BioVentrix PliCath HF Epicardial Catheter-based Ventricular Reduction (ECVR) System for left ventricular (LV) volume reduction in heart failure (HF). The System utilizes anchors that are implanted into the scarred portion of the heart, rendering the ventricle smaller.
  Other Names: Epicardial Catheter-based Ventricular Restoration; Left or Surgical Ventricular Reconstruction; Dor

SUMMARY:
The purpose of the study is to determine the safety, and feasibility of a device, which enables LV volume and radius reduction through scar exclusion in patients whose systolic HF is due to ischemic cardiomyopathy.

Appropriate subjects will have akinetic or dyskinetic scar located in the antero-septal LV distribution. Use of this device replicates the geometric reconfiguration of the ventricle achieved through surgical Left Ventricular Reconstruction (LVR), but on a beating, unsupported heart, thereby creating the option of avoiding the use of cardiopulmonary bypass pump (CBP).

DETAILED DESCRIPTION:
Congestive heart failure is the "epidemic" of cardiovascular disease (Eugene Braunwald, NEJM 1997), yet there is no cure. The American Heart Association (AHA) reports the nearly five million Americans are afflicted. Approximately 1.5 million admissions in the US are due to heart failure (HF); it is the number one cost-item for Medicare, comprising 6% of its total expenditures.

In view of the limitations of existing therapy, physicians have sought alternative treatments. In this regard, there has been longstanding interest in surgical reconstruction of the failing heart. The underlying premise has been to surgically reduce the size of the ventricular chamber by removing a portion of the ventricular wall to decrease chamber radius. A reduction of chamber radius reduces wall stress for a given pressure so that the remaining muscle is put into a more favorable mechanical state.

The BioVentrix PliCath HF System consists of implantable anchors, the delivery system, and accessories, which are sterile and biocompatible. These devices are used in the reconfiguration of the abnormal cardiac geometry that is causing dysfunction by excluding a portion of the left ventricular chamber.

The procedure is based on the premise that the beneficial effects of Left Ventricular Reconstruction (LVR) via radius and volume reduction, can be realized by excluding a portion of the scarred left ventricle wall circumference. The procedure is similar to a Dor procedure except that it utilizes a series of anchors in place of the Fontan stitch and patch to exclude infarcted tissue and reduce the size of the left ventricle chamber and the scarred left ventricle wall. Because the ventricle is not resected, it is possible to do the procedure without a cardiopulmonary bypass pump.

The validity of this concept has been documented. Geometric confirmation was initially accomplished in a bench model, where radius was decreased by 24% and volume was diminished by 35% after exclusion of an antero-septal wall segment in dilated, explanted porcine hearts.

When using the PliCath System in accomplishing LV reconfiguration, the fundamental technical maneuver is placement of a hollow needle through a predetermined site in the anterior wall scar, across the LV chamber, and through a predetermined site in the scarred interventricular septum. Once achieved, a flexible guidewire is advanced through the needle and into the free right ventricular (RV) chamber. Once the wire is completely through the septum, a dilator enables passage of a 14Fr Introducer to traverse the needle route, allowing introduction of an internal, elongated anchor which can be oriented into appropriate alignment and matched with an external anchor of identical length and alignment. The anchors, which are placed in the RV and on the epicardium as a result of the original needle passage, can be brought toward each other until contact between the two walls is established and they are apposed along their lengths. The action is repeated (i.e., repeated needle sticks and anchor placement), along the long axis of the LV until a linear portion of antero-lateral wall is in contact with a corresponding portion of the septum, excluding the entire intervening wall segment from the circumference of the chamber.

The device is designed to allow removal at any stage of deployment prior to removal of the "Leash" attached to the hinged, internal anchor.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80
* 15% ≥ LVEF ≤ 45%
* NYHA FC II-III
* 60 cc/m² ≥ LVESV/I ≤ 120 cc/m²
* Acontractile (akinetic and/or dyskinetic) scar located in the antero-septalapical region due to prior infarction as evidenced by an echocardiogram and/or an MRI
* Maintained standard medical management for at least 90 days, and at stable target (or maximum tolerated) dosages.
* Willing and competent to complete informed consent
* Viability of myocardium in regions remote from area of intended scar exclusion as evidenced by an echocardiogram and/or an MRI
* Agree to required follow-up visits

Exclusion Criteria:

* Calcified ventricular wall in the akinetic region
* Thrombus or intra-ventricular mass in left atrium or ventricle Cardiac Resynchronization Therapy (CRT) device placement within prior 60 days of enrollment
* Significant diastolic dysfunction, defined as a pseudonormal Doppler filling pattern with E/A ratio > 2
* Thin walled, paradoxically moving septal scar that would preclude successful support of the anchor pairs as evidenced by an MRI
* Cardiac valve disease which, in the opinion of the investigator, will require surgery
* Mitral Regurgitation > 1+
* Intolerance or unwillingness to take warfarin
* Functioning pacemaker leads in antero-apical RV which, in the opinion of the investigator, would interfere with anchor placement.
* Pulmonary Arterial Pressure > 60 mm Hg
* Myocardial Infarction within prior 90 days enrollment
* Previous CVA or TIA which resulted, in the opinion of the investigator, in a significant residual neurological deficit
* Co-morbid disease process with life expectancy of less than one year
* Patients with lung, kidney and/or liver transplant
* Chronic renal failure with a serum creatinine > 2 mg/dL
* Pregnant or planning to become pregnant during the study
* Enrolled in any concurrent study other than observational

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Assessment of overall rate of serious adverse device effects | 12 Months Post-operative
  The primary safety endpoint is an assessment of the overall rate of serious adverse device effects through 12 months as adjudicated by the Data Monitoring Committee.

SECONDARY OUTCOMES:
Assessment of overall rate of serious adverse events | 12 Months post-operative
  The secondary safety endpoint is an assessment of the overall rate of serious adverse events through 12 months as adjudicated by the Data Monitoring Committee.

CONTACTS AND LOCATIONS:
Locations (4):
- Pauls Stradins Hospital, Riga, Latvia
- Santariskiu Klinikus, Vilnius, Lithuania
- Jagiellonian University Hospital, Krakow, Poland
- Bakoulev Institute, Moscow, Russia

REFERENCES:
- See also: Sponsor company web site — http://www.bioventrix.com/